CLINICAL TRIAL: NCT05511714
Title: Expanded Access [11C] Methionine PET Imaging
Status: Available | Type: Expanded Access
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EXAMPT
Record Dates: First submitted 2022-08-19; First posted 2022-08-23 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Central Nervous System Tumor; Head and Neck Neoplasms
MeSH Terms: conditions — Central Nervous System Neoplasms; Head and Neck Neoplasms | interventions — Methionine; carbon-11 methionine

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: L-(11C) methionine — Injected intravenously with 20 mCi/1.7 sq m body surface area of L-[methyl-11C]methionine (maximum prescribed dose: 20 mCi).
  Other Names: methionine C 11

SUMMARY:
The participants are being asked to get this PET scan because the participants have or may have cancer in the central nervous system (head, neck, or spine), and the investigator and the patient's physician thinks that this scan may provide useful information for the participant's treatment.

Primary Objective

To provide expanded access to L-[11C]methionine as a positron-emitting tracer in children and young adults for the positron emission tomography (PET) imaging of neoplasms of the central nervous system (CNS) and head and neck to guide therapeutic management of disease.

DETAILED DESCRIPTION:
Participants receive an intravenous injection of a small (tracer) dose of L-[11C]methionine. Approximately 10 minutes later, patients undergo PET scanning to evaluate localization of the tracer.

ELIGIBILITY:
Inclusion Criteria:

* All participants under the care of a SJCRH physician with known or suspected neoplastic disease of the CNS or head and neck are eligible for participation.
* No limit on age.
* Patients of all genders and all ethnic groups under the care of a SJCRH physician.
* Female participants of child-bearing age must not be lactating due to theoretical potential harm to the infant from exposure to radiation.
* Informed consent signed by participant, parent, or guardian according to the guidelines of the Institutional Review Board.

Exclusion Criteria:

* More than six L-[11C]methionine PET scans within the previous 12 months.
* Inability or willingness of patient, parent, or guardian to consent.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Barry L. Shulkin, MD, MBA, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols